CLINICAL TRIAL: NCT06383026
Title: Understanding Breast Cancer Risk and Screening in Individuals on Hormone Therapy Through a Pilot Breast Cancer Screening Program
Brief Title: Individuals on Hormone Therapy Breast Cancer Screening Pilot
Status: Recruiting | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Chandler S Cortina, Associate Professor of Surgery, Medical College of Wisconsin
Other Study IDs: PRO00047199
Record Dates: First submitted 2024-04-17; First posted 2024-04-25 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: Mammogram; Mammography; Breast Cancer Screening; Breast Ultrasound; Breast Ultrasonography; Individuals on Hormone Therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires; Interviews as Topic; Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals on Hormone Therapy: Breast imaging data in the form of standard screening mammography in addition to screening whole breast ultrasound will be gathered and interpretations will follow the standard Breast Imaging Reporting and Data Systems.
  Insight on the perceptions and experiences of being involved in a breast cancer screening program will be gathered.
  Interventions: Diagnostic Test: Breast Cancer Screening; Other: Survey/Interview
- Breast Imaging Stakeholders: A semi-structure focus group to explore radiology faculty and staff experiences while capturing information on the perceived screening barriers, what support and/or training staff require to ensure patients are treated equitable in the screening process, and areas for providers and healthcare systems to improve breast cancer screening for individuals on hormone therapy.
  Interventions: Other: Focus Group

INTERVENTIONS:
Diagnostic Test: Breast Cancer Screening — Screening mammography as well as whole breast ultrasound interpreted by BI-RADS.
  Groups: Individuals on Hormone Therapy
Other: Survey/Interview — A mixed-methods approach including electronic surveys and one on one interviews.
  Groups: Individuals on Hormone Therapy
Other: Focus Group — A semi-structured focus group with open-ended questions that explores faculty and staff experiences in a breast cancer screening program for individuals on hormone therapy.
  Groups: Breast Imaging Stakeholders

SUMMARY:
This investigation is a prospective breast cancer screening study open to all individuals on hormone therapy. Using a mixed methods approach, the study will 1) gather prospective quantitative breast imaging data in conjunction with hormone therapy and family cancer history and 2) investigate individuals on hormone therapy perceptions and experiences in the breast cancer screening program, and 3) identify individual and systems-level barriers to breast cancer screening.

ELIGIBILITY:
Inclusion Criteria for Individuals on Hormone Therapy:

1. Males 40-75 years of age with a history of ≥9 months of estrogen and/or progesterone hormone therapy.
2. Females 40-75 years of age with any history of testosterone hormone therapy, with or without cosmetic mastectomy, but have not undergone complete mastectomy.
3. Persons who have undergone breast cancer screening before can participate.
4. Individuals who meet criteria for above eligibility and are ≥30-39 years of age with a 1st or 2nd degree family member with breast cancer.
5. Ability to speak, read, and write in English.
6. Ability to understand a written informed consent document, and the willingness to sign it.

Inclusion Criteria for Breast Radiology Faculty:

1. Board-certified radiologist that specializes in breast imaging and are an actively employed faculty member at Froedtert & the Medical College of Wisconsin (main campus location).
2. Part of the breast radiology faculty who read both ABUS and MMG of the study participants.
3. Ability to speak, read, and write in English.
4. Ability to understand a written informed consent document, and the willingness to sign it.

Inclusion Criteria for Breast Radiology Staff:

1. Must be either a technician, nurse, or clerical staff that works with the breast radiology team at Froedtert & the Medical College of Wisconsin (main campus location).
2. Ability to understand a written informed consent document, and the willingness to sign it.
3. Ability to speak, read, and write in English.

Exclusion Criteria for Individuals on Hormone Therapy

1. Females who have undergone or planned to undergo a complete mastectomy.
2. Females who are post-menopausal on estrogen +/- progesterone hormone therapy since it is a well-established risk for breast cancer).
3. A personal history of breast cancer or a known pathogenic gene mutation that increases the risk of breast cancer development (e.g., BRCA1/2, etc.) given that well-defined surveillance and screening recommendations exist for these persons.

Exclusion Criteria for Breast Radiology Faculty

1. Not a board-certified radiologist.
2. Does not specialize in breast imaging.
3. Does not read ABUS and MMG and/or has not read imaging for study participants.

Exclusion for Breast Radiology Staff

1. Does not work with the breast radiology team.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals on hormone therapy and breast cancer radiology stakeholders.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Callback and Biopsy Rates after Breast Cancer Screening | 3.5 years
  Determine the callback and biopsy rates after screening imaging of the entire individuals on hormone therapy patient cohort who complete breast imaging exams.
Reflexive Thematic Analysis of the Physical, Cognitive, and Emotional Experience of Breast Cancer Screening in Individuals on Hormone Therapy | 3.5 years
  Qualitative data utilized to identify themes around health beliefs, anxiety, and the breast cancer screening experience by describing the physical, cognitive, and emotional experience (perceived seriousness, perceived susceptibility, and anxiety) of individuals on hormone therapy cohort participants who complete surveys or participate in one-on-one interviews.
Reflexive Thematic Analysis on the Individual & System-Level Barriers to Breast Cancer Screening | 3.5 years
  Qualitative date utilized to identify individual and healthcare systems-level barriers to breast cancer screening for individuals on hormone therapy who complete surveys and/or participate in one-on-one interviews and breast imaging faculty and staff who participate in focus groups.

CONTACTS AND LOCATIONS:
Overall Officials: Chandler S Cortina, MD, MS, Principal Investigator — The Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States